CLINICAL TRIAL: NCT06592833
Title: Investigating the Role of Serotonin in the Mechanism of Action of Psilocybin in Patients With Major Depressive Disorder
Brief Title: Psilocybin With Pimavanserin Compared to Psilocybin Alone for the Treatment of Major Depressive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-23-00855
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psilocybin; pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin + Pimavanserin (Active Comparator): single dose Psilocybin and single dose Pimavanserin
  Interventions: Drug: Psilocybin; Drug: Pimavanserin
- Psilocybin + Placebo (Placebo Comparator): single dose Psilocybin and single dose Placebo
  Interventions: Drug: Psilocybin; Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — Psilocybin, 25mg, given once orally.
Drug: Pimavanserin — Pimavanserin, 34mg, given once orally
  Other Names: Nuplazid
  Arms: Psilocybin + Pimavanserin
Drug: Placebo — Matching placebo.
  Arms: Psilocybin + Placebo

SUMMARY:
This is an interventional, parallel arm assignment treatment study in individuals with Major Depressive Disorder (MDD). Each individual will be treated with a single dose of pimavanserin or placebo plus a single dose of psilocybin. Evaluations will be taken before dosing and following dosing at several timepoints up to 5 weeks post-dosing.

DETAILED DESCRIPTION:
In this study, the researchers want to probe the role of the 5-HT2A receptor in mediating the subjective effects of psilocybin. While previous studies have shown that blockage of the 5-HT2A receptor reduces the psychedelic experience in humans, an animal study revealed that blockage of the 5- HT2A receptor abolished the psychedelic effects without affecting the antidepressant response. This suggests that the pathway responsible for the antidepressant response is dissociated from the psychedelic experience pathway, which is mediated by 5-HT2A signaling.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 years, any gender
* Current primary diagnosis of Unipolar Major Depressive Disorder (MDD) without psychotic features using DSM-5 criteria
* 24-item Hamilton Rating Scale for Depression (HRSD) ≥16
* Current diagnosis of Major Depressive Episode (MDE)
* Capable of providing informed consent and complying with study procedures
* Currently using or agreeing to use a highly effective contraception, if person of childbearing potential (such as condoms, IUD, or oral contraceptive), for duration of the study. Male participants agree to use highly effective contraception with partners of childbearing potential
* Discontinuation of any serotonergic drug for at least 2 weeks or 5 half-lives (whichever of the two is longer) prior to psilocybin exposure

Exclusion Criteria:

* Any severity of substance use disorder in the last 6 months (excluding tobacco use disorder) as determined by DSM-V criteria via the SCID
* Current psychiatric hospitalization or psychiatric hospitalization within the last 6 months
* Use of psychedelics in the last 12 months
* Non-medical or illicit use of ketamine in the past 12 months
* Negative reaction after prior use of psychedelics
* Past or current psychotic disorder (including psychotic MDD), mania, or bipolar disorder
* Severe depression as indicated by Clinical Global Impressions (CGI)-Severity score ≥ 5 at baseline
* Significant suicidal ideation as indicated by C-SSRS > 2 in the past 6 months at time of screening
* Suicide attempt in the past 2 years, or clinician concern that the patient poses a risk to self or others
* Acute, severe, or unstable medical illness
* Weight > 300 lbs., or girth size incompatible with scanner bore
* Any conditions/qualities that make participation in MRI imaging unsafe*
* Any physical or intellectual disability adversely affecting ability to complete assessments.
* Current pregnancy or currently breast feeding.
* Any clinically significant abnormal lab test result, including clinically significant abnormal baseline liver and/or renal function tests
* Currently being treated with a contraindicated medication. Contraindicated medications include antipsychotic medications, serotonergic antidepressant medications, and mood stabilizers that may attenuate the effects of psilocybin. Strong CYP3A4 inhibitors and inducers are also contraindicated. UGT1A9 and UGT1A10 inhibitors, monoamine oxidase, and aldehyde or alcohol dehydrogenase inhibitors are prohibited concomitant medications.
* History of abnormal QT prolongation or QTc interval >450 ms on screening
* Use of medications known to prolong the QT interval
* Any congenital prolongation of the QT interval or a family history of long QT syndrome
* A family history of sudden cardiac or unexplained death
* A family history in a first-degree relative of psychosis/schizophrenia or related disorders
* A first-degree family history of bipolar disorder
* A history of cardiac arrhythmias or who require treatment with an antiarrhythmic medication
* A history of any cardiovascular disorder/condition known to increase the possibility of QT prolongation, or any other risk factors for prolonged QT interval/tosades de pointes (including symptomatic bradycardia, hypokalemia, hypomagnesemia, hypocalcemia, heart failure, or Brugada Syndrome)
* Preexisting cardiovascular conditions, including cardiac valvulopathy, pulmonary hypertension, hypertension, tachycardia, and any cardiovascular conditions that may be worsened/exacerbated by elevated blood pressure or heart rate.
* Baseline vital sign parameters at screening and on day of dosing prior to dose that exceed to the following values for systolic blood pressure (SBP), diastolic (DBP), and heart rate (HR): SBP > 139 mmHg, DBP 89 mmHg, and HR > 90 bpm
* Hypersensitivity to either psilocybin or pimavanserin
* Psychiatric or other condition judged to be incompatible with establishment of rapport with therapy team and/or safe exposure to psilocybin
* Positive urine toxicology at screening
* Any clinically significant abnormalities on 12-lead electrocardiogram (ECG)
* Mini-Mental State Examination (MMSE) score < 25
* Brief Psychiatric Rating Scale (BPRS-6) > 5
* Potential fall risk

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Mystical Experience Questionnaire (MEQ-30) Score | 6 hours post-treatment
  Acute subjective effects of psilocybin measured by the Mystical Experience Questionnaire (MEQ-30). Full Scale ranges from 0 to 150, with higher scores indicating more mystical experience.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) Score | 7 days after dosing
  The Montgomery-Åsberg Depression Rating Scale (MADRS) will be used to measure improvement in depressive symptoms 7 days after dosing. This 10-item clinician-rated scale measures the severity of depressive symptoms. Full scale ranges from 0 to 60, with higher scores indicating more depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, Principal Investigator — Icahn School of Medicine at Mount Sinai; Rachel Fremont, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, Center for Psychedelic Therapy Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Because this study is privately funded, the research team is not required to share IPD.